CLINICAL TRIAL: NCT00034125
Title: a Phase 3 Randomized Double Blind Evaluation of LY353381 Compared With Tamoxifen in Women With Locally Advanced or Metastatic Breast Cancer.
Brief Title: Phase 3 Study of LY353381 Vs Tamoxifen in Women With Locally Advanced or Metastatic Breast Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3883; H4Z-MC-JWXD
Record Dates: First submitted 2002-04-23; First posted 2002-04-24 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Breast Neoplasms
Keywords: cancer; metastatic breast cancer; hormonal therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — LY 353381; Tamoxifen

INTERVENTIONS:
Drug: LY353381
Drug: tamoxifen

SUMMARY:
To determine the safety and efficacy of LY353381 when compared to tamoxifen in women with advanced or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria

1. Locally advanced or metastatic breast cancer
2. Bi-dimensionally measurable disease

Exclusion Criteria

1. Prior hormonal therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (11):
- United States (4):
  - Miami, Florida
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Nashville, Tennessee
- Argentina (2):
  - Capital Federal, Buenos Aires
  - Ciudad de Buenos Aires, Buenos Aires F.D.
- Chile (2):
  - Las Condes, Santiago Metropolitan
  - Providencia, Santiago Metropolitan
- Ahmedabab, Gujarat, India
- Mexico (2):
  - Mexico City, Benito Juarez
  - Colima, Colima